CLINICAL TRIAL: NCT02353663
Title: Rheumatic Heart Disease in Peru: Prevalence and Cardiovascular Outcomes Among Schoolchildren
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Instituto de Cardiología Paredes-Horna, Arequipa (Unknown); Hospital Nacional Carlos Alberto Seguin Escobedo - EsSalud (Other)
Responsible Party: Sponsor
Other Study IDs: 1927-CIEI_USMP-CCM
Record Dates: First submitted 2015-01-28; First posted 2015-02-03 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatic Heart Disease; Acute Rheumatic Fever
Keywords: Rheumatic heart disease; Rheumatic fever; Mitral regurgitation; Aortic regurgitation; Mitral stenosis
MeSH Terms: conditions — Rheumatic Heart Disease; Rheumatic Fever; Mitral Valve Insufficiency; Aortic Valve Insufficiency; Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: Schoolgoing children 5 to 16 years of age
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Echocardiography examination

SUMMARY:
Rheumatic heart disease remains a major challenge in low and middle income countries. Early detection of clinically silent valvular lesions by screening echocardiography allows timely implementation of secondary antibiotic prevention, and may prevent progression of disease to severe valvular damage and heart failure. The objective of the study is to assess the prevalence of rheumatic heart disease among schoolchildren in Arequipa, Peru. Subsequently, the investigators will evaluate progression of disease in children with early stages of subclinical rheumatic heart disease.

The investigators will perform a population-based observational survey for rheumatic heart disease using portable echocardiography among schoolchildren aged 5 to 16 years from randomly selected public and private schools. Rheumatic heart disease will be documented both according to the modified World Health Organization definition and the echocardiographic criteria suggested by the World Heart Federation.

DETAILED DESCRIPTION:
Background

Rheumatic fever complicated by rheumatic heart disease continues to be a major contributor to morbidity and premature death in low- and middle-income countries where it accounts for up to a quarter of a million deaths every year. Rheumatic fever results from an autoimmune response to groups A streptococcal pharyngitis and may progress to rheumatic heart disease with cumulative exposure. Data on prevalence of rheumatic heart disease in Latin America is scarce and ranges from 1.3/1000 as assessed by cardiac auscultation to 4.1/1000 as assessed by echocardiography.

Secondary antibiotic prevention and inclusion of patients with rheumatic heart disease in a registry with close follow-up has been demonstrated to reduce the cardiovascular sequelae associated with disease progression.

The natural course of early, clinically silent stages of rheumatic heart disease is largely unknown. Disease regression has been reported in up to one third of children with early morphological valvular changes consistent with rheumatic heart disease.

Objective

The objective of the study is to assess the prevalence of rheumatic heart disease among schoolchildren in Arequipa, Peru. Subsequently, the investigators will investigate progression of disease in children with early stages of subclinical rheumatic heart disease.

Methods

The investigators will perform a population-based observational survey for rheumatic heart disease using portable echocardiography among schoolchildren aged 5 to 16 years from randomly selected public and private schools. Rheumatic heart disease will be documented both according to the modified World Health Organization definition and the echocardiographic criteria suggested by the World Heart Federation. Children diagnosed with rheumatic heart disease will be started on secondary antibiotic prevention and included into a prospective registry with longitudinal follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren aged 5 to 15 years
* Written informed consent

Exclusion Criteria

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Schoolchildren aged 5 to 16 years from Arequipa,Peru. Among 457 schools we randomly selected 40 classes from 20 schools using a mutlistage sampling strategy.
Sampling Method: Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Rheumatic heart disease according to WHO and WHF criteria | 12 months

SECONDARY OUTCOMES:
Progression of disease | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, MD, Principal Investigator — Bern University Hospital
Locations (2):
- Instituto de Cardiología Paredes-Horna, Arequipa, Arequipa, Peru
- Department of Cardiology, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Rothenbuhler M, O'Sullivan CJ, Stortecky S, Stefanini GG, Spitzer E, Estill J, Shrestha NR, Keiser O, Juni P, Pilgrim T. Active surveillance for rheumatic heart disease in endemic regions: a systematic review and meta-analysis of prevalence among children and adolescents. Lancet Glob Health. 2014 Dec;2(12):e717-26. doi: 10.1016/S2214-109X(14)70310-9. PMID 25433627
- [Background] Carapetis JR, Steer AC, Mulholland EK, Weber M. The global burden of group A streptococcal diseases. Lancet Infect Dis. 2005 Nov;5(11):685-94. doi: 10.1016/S1473-3099(05)70267-X. PMID 16253886
- [Background] Pelajo CF, Lopez-Benitez JM, Torres JM, de Oliveira SK. Adherence to secondary prophylaxis and disease recurrence in 536 Brazilian children with rheumatic fever. Pediatr Rheumatol Online J. 2010 Jul 26;8:22. doi: 10.1186/1546-0096-8-22. PMID 20659324
- [Derived] Bartkowiak J, Spitzer E, Kurmann R, Zurcher F, Krahenmann P, Garcia-Ruiz V, Mercado J, Ryffel C, Losdat S, Llerena N, Torres P, Lanz J, Stocker M, Ren B, Glockler M, Pilgrim T. The impact of obesity on left ventricular hypertrophy and diastolic dysfunction in children and adolescents. Sci Rep. 2021 Jun 22;11(1):13022. doi: 10.1038/s41598-021-92463-x. PMID 34158575
- [Derived] Spitzer E, Mercado J, Islas F, Rothenbuhler M, Kurmann R, Zurcher F, Krahenmann P, Llerena N, Juni P, Torres P, Pilgrim T. Screening for Rheumatic Heart Disease among Peruvian Children: A Two-Stage Sampling Observational Study. PLoS One. 2015 Jul 24;10(7):e0133004. doi: 10.1371/journal.pone.0133004. eCollection 2015. PMID 26208006